CLINICAL TRIAL: NCT05122832
Title: Preventive and Personalized Medicine (2021-2023)
Brief Title: Prevalence of NCD Risk Factors in Kazakhstan
Status: Completed | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Head of the Laboratory of Experimental Medicine, Asfendiyarov Kazakh National Medical University
Other Study IDs: 1197
Record Dates: First submitted 2021-09-29; First posted 2021-11-17 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Non-Communicable Chronic Diseases
MeSH Terms: conditions — Noncommunicable Diseases | interventions — Hematologic Tests; Spirometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study Group: Population of Kazakhstan
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: STEPwise Approach to NCD Risk Factor Surveillance (STEPS); Diagnostic Test: Spirometry

INTERVENTIONS:
Diagnostic Test: Blood test — Glucose Glycosylated hemoglobin Triglycerides Total cholesterol HDL Cholesterol LDL Cholesterol Creatinine COVID-19 Antibody IgM to N protein SARS-Cov-2 (Abbott) COVID-19 Antibody IgG to N protein SARS-Cov-2 (Abbott)
Diagnostic Test: STEPwise Approach to NCD Risk Factor Surveillance (STEPS) — The WHO STEPwise Approach to NCD Risk Factor Surveillance (STEPS) is a simple, standardized method for collecting, analysing and disseminating data on key NCD risk factors in countries. The survey instrument covers key behavioral risk factors: tobacco use, alcohol consumption, physical activity, unhealthy diet, as well as key biological risk factors: overweight and obesity, raised blood pressure, raised blood glucose, and abnormal blood lipids. Through the use of expanded modules, the survey instrument can be expanded to cover a range of topics beyond these risk factors, such as oral health, sexual health and road safety.
Diagnostic Test: Spirometry — Spirometry is a common office test used to assess how well your lungs work by measuring how much air you inhale, how much you exhale and how quickly you exhale.

SUMMARY:
This is a cross-sectional study that aims to study the prevalence of risk factors of noncommunicable diseases in people aged 18 to 69 years using the standardized and adopted STEPS questionnaire in the Republic of Kazakhstan.

DETAILED DESCRIPTION:
The WHO STEPwise Approach to NCD Risk Factor Surveillance (STEPS) is a simple, standardized method for collecting, analysing and disseminating data on key NCD risk factors in countries. The survey instrument covers key behavioral risk factors: tobacco use, alcohol consumption, physical activity, unhealthy diet, as well as key biological risk factors: overweight and obesity, raised blood pressure, raised blood glucose, and abnormal blood lipids.

ELIGIBILITY:
Inclusion Criteria:

* Age Limits 18-69 years

Ages: 18 Years to 69 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All ethnic groups in Kazakhstan
Sampling Method: Probability Sample
Enrollment: 20400 (Actual)
Dates: Start 2021-10-23 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
tobacco use | 1 year
  currently smoke tobacco, currently smoke tobacco daily, age started smoking, daily smokers smoking manufactured cigarettes
alcohol consumption | 1 year
  lifetime abstainers, past 12 month abstainers, currently drink (drank alcohol in the past 30 days), heavy episodic drinking (6 or more drinks on any occasion in the past 30 days).
physical activity | 1 year
  insufficient physical activity (defined as < 150 minutes of moderate-intensity activity per week, or equivalent), physical activity on average per day (minutes), not engaging in vigorous activity.
unhealthy diet | 1 year
  days fruit consumed in a typical week, servings of fruit consumed on average per day, days vegetables consumed in a typical week, servings of vegetables consumed on average per day, less than 5 servings of fruit and/or vegetables on average per day, always or often add salt or salty sauce to their food before eating or as they are eating, always or often eat processed foods high in salt.
BMI | 1 year
  overweight (BMI ≥ 25 kg/m2), obese (BMI ≥ 30 kg/m2), normal weight
raised blood pressure | 1 year
  systolic blood pressure - SBP (mmHg), including those currently on medication for raised BP, diastolic blood pressure - DBP (mmHg), including those currently on medication for raised BP, raised BP (SBP ≥ 140 and/or DBP ≥ 90 mmHg or currently on medication for raised BP), raised BP (SBP ≥ 140 and/or DBP ≥ 90 mmHg or currently on medication for raised BP) who are not currently on medication for raised BP.
raised blood glucose | 1 year
  fasting blood glucose, including those currently on medication for raised blood glucose, impaired fasting glycaemia (plasma venous value ≥6.1 mmol/L (110 mg/dl) and <7.0 mmol/L (126 mg/dl)), raised fasting blood glucose (plasma venous value ≥ 7.0 mmol/L (126 mg/dl)) or currently on medication for raised blood glucose.
abnormal blood lipids | 1 year
  total blood cholesterol, including those currently on medication for raised cholesterol, raised total cholesterol,

CONTACTS AND LOCATIONS:
Overall Officials: Timur M Saliev, Principal Investigator — S.D. Asfendiyarov Kazakh National Medical University; Ildar Fakhradiyev, PhD, Study Chair — S.D. Asfendiyarov Kazakh National Medical University; Mukhtar B Kulimbet, MD/MSc, Study Director — S.D. Asfendiyarov Kazakh National Medical University; Zhumaly A Kauyzbay, PhD, AP, Principal Investigator — Joint Stock Company - South Kazakhstan Medical Academy; Samat S Saparbayev, PhD, Principal Investigator — West Kazakhstan Marat Ospanov Medical University; Alma U Nurtazina, MD/PhD, Principal Investigator — NCJSC Semey Medical University; Bayan A Ainabekova, MD/DMSc, Principal Investigator — NCJSC Astana Medical University; Anar A Turmukhambetova, DMSc, Principal Investigator — NCJSC Karaganda Medical University; Maksut K Kulzhanov, DMSc, Principal Investigator — Kazakhstan's Medical University "KSPH"
Locations (1):
- Kazakhstan, Almaty, Kazakhstan

REFERENCES:
- [Derived] Baspakova A, Abitova AZ, Mussin NM, Kaliyev AA, Yerimbetova G, Zhumagaliyeva S, Ashimova Z, Zhilisbayeva KR, Umbetova AA, Nurtazina AU, Tamadon A. Sex differentials in the prevalence of behavioral risk factors and non-communicable diseases in adult populations of West Kazakhstan. Front Public Health. 2024 Feb 14;12:1333887. doi: 10.3389/fpubh.2024.1333887. eCollection 2024. PMID 38420037
- [Derived] Nursultanova L, Kabulbayev K, Ospanova D, Tazhiyeva A, Datkhayev U, Saliev T, Tanabayeva S, Fakhradiyev I. Prevalence of chronic kidney disease in Kazakhstan: evidence from a national cross-sectional study. Sci Rep. 2023 Sep 7;13(1):14710. doi: 10.1038/s41598-023-42031-2. PMID 37679536